CLINICAL TRIAL: NCT03706768
Title: Degradation of the Glycocalyx in Delayed Cerebral Ischemia After Aneurysmal Subarachnoid Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Danny Theodore, MD, Assistant Professor of Anesthesiology, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 170016
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Intervention Model Description: Aneurysmal Subarachnoid Hemorrhage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glycocalyx (Other): degree of glycocalyx breakdown in patients with aSAH
  Interventions: Other: Glycocalyx

INTERVENTIONS:
Other: Glycocalyx — Measure Degradation of the Glycocalyx

SUMMARY:
This study will provide novel information to the literature base for the pathophysiology of aneurysmal subarachnoid hemorrhage. The association of breakdown products in the serum of aSAH patients were reported in a very small case series of 3 patients, as mentioned above. However, while their results are intriguing and encouraging, our study will provide more definitive information about the GC in aSAH. If there is a positive correlation, the results of this study will guide future investigations into new therapies for this devastating disease such as MMP inhibition with doxycycline.

DETAILED DESCRIPTION:
1. The study will aim to recruit all eligible patients at UTMCK and the University of Virginia hospital over a 12 month period. Our main outcome measure is degradation of the glycocalyx in patients with aSAH. All eligible patients with confirmed aSAH admitted to the neuro-intensive care unit will be enrolled after consent is obtained from the family and/or the patient. Serum samples will be drawn from each patient on admission (day 1) and every other day until day 13 for a total of 7 samples per patient.

   The following serum tests will be performed:
2. Measurement of serum syndecan-1 by ELISA
3. Measurement of serum heparan-sulfate by ELISA
4. Measurement of serum matrix metalloproteinases -9
5. Measurement of serum matrix-metalloproteinase-1
6. Measurement of urinary microalbumin-to-creatinine ratio
7. Measurement of daily TCDs (all patients currently receive daily TCDs as part of the aSAH protocol at UTMCK and UVA Hospital)
8. Outcomes:

   a) Chart review: i) Incidence of DCI as defined by a consensus committee on this subject and published in the journal Stroke [29].

   ii) In-hospital mortality will be recorded b) Follow-up performed by phone call or searching the Social Security Death Index [30]: i) 30-day mortality ii) 90-day mortality c) Outcomes follow-up: i) The Glasgow Outcome Scale 12 weeks post aSAH [31]

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 years of age and older

  * Cerebral aneurysm on CT-angio

Exclusion Criteria:

* • comfort care only orders,

  * the absence of an aneurysm on CT-angiography,
  * onset of aneurysm rupture > 24 hours,
  * and inability to obtain informed consent from patient or family pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Syndecan-1 and heparin sulfate | day 0 through day 13
  Compare the degree of glycocalyx breakdown in patients with aSAH who develop delayed cerebral ischemia (DCI) to those that do not develop DCI. This will be completed by measuring the breakdown of Syndecan-1 and heparin sulfate in the blood.

SECONDARY OUTCOMES:
serum Matrix metalloproteinase-1 and Matrix metalloproteinase-9 | day 0 through day 13
  serum MMP-9 and MMP-1 will be levels will be measured as serum MMP concentrations have been positively correlated with the incidence of delayed cerebral ishemia
urinary microalbumin-to-creatinine ratio (MACR) | day 0 through day13
  urinary microalbumin-to-creatinine ratio (MACR) will be measured as it is marker of systemic damage to the glycocalyx

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Theodore, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bogason ET, Anderson B, Brandmeir NJ, Church EW, Cooke J, Davies GM, Hussain N, Patel AS, Payne R, Rohatgi P, Sieg E, Zalatimo O, Ziu E. The epidemiology of admissions of nontraumatic subarachnoid hemorrhage in the United States. Neurosurgery. 2014 Feb;74(2):227-9. doi: 10.1227/NEU.0000000000000240. No abstract available. PMID 24435139
- [Background] Macdonald RL, Higashida RT, Keller E, Mayer SA, Molyneux A, Raabe A, Vajkoczy P, Wanke I, Bach D, Frey A, Marr A, Roux S, Kassell N. Clazosentan, an endothelin receptor antagonist, in patients with aneurysmal subarachnoid haemorrhage undergoing surgical clipping: a randomised, double-blind, placebo-controlled phase 3 trial (CONSCIOUS-2). Lancet Neurol. 2011 Jul;10(7):618-25. doi: 10.1016/S1474-4422(11)70108-9. Epub 2011 Jun 2. PMID 21640651
- [Background] Rowland MJ, Hadjipavlou G, Kelly M, Westbrook J, Pattinson KT. Delayed cerebral ischaemia after subarachnoid haemorrhage: looking beyond vasospasm. Br J Anaesth. 2012 Sep;109(3):315-29. doi: 10.1093/bja/aes264. PMID 22879655
- [Background] Collins SR, Blank RS, Deatherage LS, Dull RO. Special article: the endothelial glycocalyx: emerging concepts in pulmonary edema and acute lung injury. Anesth Analg. 2013 Sep;117(3):664-674. doi: 10.1213/ANE.0b013e3182975b85. Epub 2013 Jul 8. PMID 23835455
- [Background] Alphonsus CS, Rodseth RN. The endothelial glycocalyx: a review of the vascular barrier. Anaesthesia. 2014 Jul;69(7):777-84. doi: 10.1111/anae.12661. Epub 2014 Apr 28. PMID 24773303
- [Background] Yang Y, Schmidt EP. The endothelial glycocalyx: an important regulator of the pulmonary vascular barrier. Tissue Barriers. 2013 Jan 1;1(1):e23494. doi: 10.4161/tisb.23494. PMID 24073386
- [Background] Singh A, Ramnath RD, Foster RR, Wylie EC, Friden V, Dasgupta I, Haraldsson B, Welsh GI, Mathieson PW, Satchell SC. Reactive oxygen species modulate the barrier function of the human glomerular endothelial glycocalyx. PLoS One. 2013;8(2):e55852. doi: 10.1371/journal.pone.0055852. Epub 2013 Feb 14. PMID 23457483
- [Background] Ince C, Mayeux PR, Nguyen T, Gomez H, Kellum JA, Ospina-Tascon GA, Hernandez G, Murray P, De Backer D; ADQI XIV Workgroup. THE ENDOTHELIUM IN SEPSIS. Shock. 2016 Mar;45(3):259-70. doi: 10.1097/SHK.0000000000000473. PMID 26871664
- [Background] Bell JD, Rhind SG, Di Battista AP, Macdonald RL, Baker AJ. Biomarkers of Glycocalyx Injury are Associated with Delayed Cerebral Ischemia Following Aneurysmal Subarachnoid Hemorrhage: A Case Series Supporting a New Hypothesis. Neurocrit Care. 2017 Jun;26(3):339-347. doi: 10.1007/s12028-016-0357-4. PMID 28000132
- [Background] Becker BF, Jacob M, Leipert S, Salmon AH, Chappell D. Degradation of the endothelial glycocalyx in clinical settings: searching for the sheddases. Br J Clin Pharmacol. 2015 Sep;80(3):389-402. doi: 10.1111/bcp.12629. Epub 2015 May 22. PMID 25778676
- [Background] Lipowsky HH. The endothelial glycocalyx as a barrier to leukocyte adhesion and its mediation by extracellular proteases. Ann Biomed Eng. 2012 Apr;40(4):840-8. doi: 10.1007/s10439-011-0427-x. Epub 2011 Oct 8. PMID 21984514
- [Background] Triglia T, Mezzapesa A, Martin JC, Verdier M, Lagier D, Dufour H, Bruder N, Alessi MC, Velly LJ. Early matrix metalloproteinase-9 concentration in the first 48 h after aneurysmal subarachnoid haemorrhage predicts delayed cerebral ischaemia: An observational study. Eur J Anaesthesiol. 2016 Sep;33(9):662-9. doi: 10.1097/EJA.0000000000000494. PMID 27355865
- [Background] Tromp J, van der Pol A, Klip IT, de Boer RA, Jaarsma T, van Gilst WH, Voors AA, van Veldhuisen DJ, van der Meer P. Fibrosis marker syndecan-1 and outcome in patients with heart failure with reduced and preserved ejection fraction. Circ Heart Fail. 2014 May;7(3):457-62. doi: 10.1161/CIRCHEARTFAILURE.113.000846. Epub 2014 Mar 19. PMID 24647119
- [Background] Neves FM, Meneses GC, Sousa NE, Menezes RR, Parahyba MC, Martins AM, Liborio AB. Syndecan-1 in Acute Decompensated Heart Failure--Association With Renal Function and Mortality. Circ J. 2015;79(7):1511-9. doi: 10.1253/circj.CJ-14-1195. Epub 2015 Apr 17. PMID 25891890
- [Background] Ostrowski SR, Gaini S, Pedersen C, Johansson PI. Sympathoadrenal activation and endothelial damage in patients with varying degrees of acute infectious disease: an observational study. J Crit Care. 2015 Feb;30(1):90-6. doi: 10.1016/j.jcrc.2014.10.006. Epub 2014 Oct 8. PMID 25457118
- [Background] Chelazzi C, Villa G, Mancinelli P, De Gaudio AR, Adembri C. Glycocalyx and sepsis-induced alterations in vascular permeability. Crit Care. 2015 Jan 28;19(1):26. doi: 10.1186/s13054-015-0741-z. PMID 25887223
- [Background] Dull RO, Cluff M, Kingston J, Hill D, Chen H, Hoehne S, Malleske DT, Kaur R. Lung heparan sulfates modulate K(fc) during increased vascular pressure: evidence for glycocalyx-mediated mechanotransduction. Am J Physiol Lung Cell Mol Physiol. 2012 May 1;302(9):L816-28. doi: 10.1152/ajplung.00080.2011. Epub 2011 Dec 9. PMID 22160307
- [Background] Nieuwdorp M, van Haeften TW, Gouverneur MC, Mooij HL, van Lieshout MH, Levi M, Meijers JC, Holleman F, Hoekstra JB, Vink H, Kastelein JJ, Stroes ES. Loss of endothelial glycocalyx during acute hyperglycemia coincides with endothelial dysfunction and coagulation activation in vivo. Diabetes. 2006 Feb;55(2):480-6. doi: 10.2337/diabetes.55.02.06.db05-1103. PMID 16443784
- [Background] Fischer M, Dietmann A, Beer R, Broessner G, Helbok R, Pfausler B, Schmutzhard E, Lackner P. Differential regulation of matrix-metalloproteinases and their tissue inhibitors in patients with aneurysmal subarachnoid hemorrhage. PLoS One. 2013;8(3):e59952. doi: 10.1371/journal.pone.0059952. Epub 2013 Mar 28. PMID 23555845
- [Background] Satoh M, Date I, Ohmoto T, Perkins E, Parent AD. The expression and activation of matrix metalloproteinase-1 after subarachnoid haemorrhage in rats. Acta Neurochir (Wien). 2005 Feb;147(2):187-92; discussion 192-3. doi: 10.1007/s00701-004-0435-9. PMID 15605197
- [Background] Endo K, Takino T, Miyamori H, Kinsen H, Yoshizaki T, Furukawa M, Sato H. Cleavage of syndecan-1 by membrane type matrix metalloproteinase-1 stimulates cell migration. J Biol Chem. 2003 Oct 17;278(42):40764-70. doi: 10.1074/jbc.M306736200. Epub 2003 Aug 6. PMID 12904296
- [Background] Terao Y, Takada M, Tanabe T, Ando Y, Fukusaki M, Sumikawa K. Microalbuminuria is a prognostic predictor in aneurysmal subarachnoid hemorrhage. Intensive Care Med. 2007 Jun;33(6):1000-6. doi: 10.1007/s00134-007-0617-z. Epub 2007 Mar 27. PMID 17387450
- [Background] Salmon AH, Satchell SC. Endothelial glycocalyx dysfunction in disease: albuminuria and increased microvascular permeability. J Pathol. 2012 Mar;226(4):562-74. doi: 10.1002/path.3964. PMID 22102407
- [Background] Lee H, Park JW, Kim SP, Lo EH, Lee SR. Doxycycline inhibits matrix metalloproteinase-9 and laminin degradation after transient global cerebral ischemia. Neurobiol Dis. 2009 May;34(2):189-98. doi: 10.1016/j.nbd.2008.12.012. Epub 2009 Jan 6. PMID 19200854
- [Background] Pires PW, Rogers CT, McClain JL, Garver HS, Fink GD, Dorrance AM. Doxycycline, a matrix metalloprotease inhibitor, reduces vascular remodeling and damage after cerebral ischemia in stroke-prone spontaneously hypertensive rats. Am J Physiol Heart Circ Physiol. 2011 Jul;301(1):H87-97. doi: 10.1152/ajpheart.01206.2010. Epub 2011 May 6. PMID 21551278
- [Background] Cerisano G, Buonamici P, Valenti R, Sciagra R, Raspanti S, Santini A, Carrabba N, Dovellini EV, Romito R, Pupi A, Colonna P, Antoniucci D. Early short-term doxycycline therapy in patients with acute myocardial infarction and left ventricular dysfunction to prevent the ominous progression to adverse remodelling: the TIPTOP trial. Eur Heart J. 2014 Jan;35(3):184-91. doi: 10.1093/eurheartj/eht420. Epub 2013 Oct 8. PMID 24104875
- [Background] Li C, Li X, Shen Q, Li Y, He L, Li M, Tang Y, Wang Y, He Q, Peng Y. Critical role of matrix metalloproteinase-9 in acute cold exposure-induced stroke in renovascular hypertensive rats. J Stroke Cerebrovasc Dis. 2013 Nov;22(8):e477-85. doi: 10.1016/j.jstrokecerebrovasdis.2013.05.016. Epub 2013 Jun 22. PMID 23800500
- [Background] Chaudhry K, Rogers R, Guo M, Lai Q, Goel G, Liebelt B, Ji X, Curry A, Carranza A, Jimenez DF, Ding Y. Matrix metalloproteinase-9 (MMP-9) expression and extracellular signal-regulated kinase 1 and 2 (ERK1/2) activation in exercise-reduced neuronal apoptosis after stroke. Neurosci Lett. 2010 Apr 26;474(2):109-14. doi: 10.1016/j.neulet.2010.03.020. Epub 2010 Mar 16. PMID 20298757